CLINICAL TRIAL: NCT04276805
Title: Non-invasive Nerve Stimulation and Cognitive Training to Improve Cognitive Performance in Healthy Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB201902991
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Aging
MeSH Terms: interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- tVNS group (Active Comparator): Participants will undergo cognitive training with tVNS
  Interventions: Device: Transcutaneous vagal nerve stimulation (tVNS); Behavioral: cognitive training
- Sham group (Sham Comparator): Participants will undergo cognitive training with earlobe sham
  Interventions: Behavioral: cognitive training

INTERVENTIONS:
Device: Transcutaneous vagal nerve stimulation (tVNS) — a non-invasive and safe technique that transiently enhances brain GABA and noradrenaline levels.
  Arms: tVNS group
Behavioral: cognitive training — A program of regular mental activities purported to maintain or improve one's cognitive abilities.

SUMMARY:
We need better tools to both enhance brain health and improve cognitive performance in healthy brain aging so that it can be delayed, reduced, or even reversed. The present proposal is designed to evaluate the pairing of cognitive training with a non-invasive neurostimulation technology that has shown promise in both increasing neuroplasticity and in enhancing cognitive performance, transcutaneous vagal nerve stimulation (tVNS).

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals willing to commit to study requirements

Exclusion Criteria:

* Neurological disorders to include traumatic brain injury.
* Evidence of dementia .
* Major psychiatric illness
* Unstable and chronic medical conditions.
* MRI contraindications (e.g., pregnancy, claustrophobia, metal implants that are contraindicated for MRI).
* Physical impairment precluding motor response or lying still or walking
* Hearing or vision deficits that will not allow for completion of assessments

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in working memory and processing speed contributors | Baseline to 2 weeks
  The Posit Science BrainHQ

CONTACTS AND LOCATIONS:
Overall Officials: John Williamson, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Arizona, Tucson, Arizona
  - University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No